CLINICAL TRIAL: NCT07085520
Title: A Clinical Study Evaluating the Dermal Safety of Soluble Denosumab Microneedle Patches
Acronym: CSEDSSDMP
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20250379
Record Dates: First submitted 2025-06-12; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis; Osteoarthritis (OA) of the Knee; Osteoporosis; Osteoporosis (Senile); Healthy
MeSH Terms: conditions — Osteoarthritis; Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Microneedle with Saline (Placebo Comparator): This study arm uses microneedle patches loaded with saline as a control to assess the skin safety of the microneedle patches. Participants will apply 4 microneedle patches around their knee and avoid behaviors that may affect skin condition during the study.
  Interventions: Drug: Saline Microneedle Patch
- Microneedle with 0.24mg Denosumab (Experimental): This study arm uses microneedle patches loaded with 0.24mg of denosumab to evaluate the skin safety and tolerability of the microneedle patch. Participants will apply 4 microneedle patches around their knee and avoid behaviors that may affect skin condition during the study.
  Interventions: Drug: Microneedle with 0.24mg Denosumab
- Microneedle with 1.2mg Denosumab (Experimental): This study arm uses microneedle patches loaded with 1.2mg of denosumab to evaluate the skin safety and tolerability of the microneedle patch. Participants will apply 4 microneedle patches around their knee and avoid behaviors that may affect skin condition during the study.
  Interventions: Drug: Microneedle with 1.2mg Denosumab
- Microneedle with 6mg Denosumab (Experimental): This study arm uses microneedle patches loaded with 6mg of denosumab to evaluate the skin safety and tolerability of the microneedle patch. Participants will apply 4 microneedle patches around their knee and avoid behaviors that may affect skin condition during the study.
  Interventions: Drug: Microneedle with 6mg Denosumab

INTERVENTIONS:
Drug: Microneedle with 0.24mg Denosumab — This intervention uses microneedle patches loaded with 0.24mg of denosumab. The patch is made of a biocompatible material, polyvinyl pyrrolidone (PVP), and is applied to the skin around the knee. It aims to evaluate the skin safety and tolerability of the microneedle patch at this specific dose. Participants will apply 4 microneedle patches around their knee and avoid behaviors that may affect skin condition during the study.
  Other Names: Soluble Denosumab Microneedle Patch
  Arms: Microneedle with 0.24mg Denosumab
Drug: Saline Microneedle Patch — This intervention involves the use of a microneedle patch loaded with saline. The patch is made of a biocompatible material, polyvinyl pyrrolidone (PVP), and is applied to the skin around the knee. It serves as a control to assess the skin safety of the microneedle patch without the active drug. Participants will apply 4 microneedle patches around their knee and avoid behaviors that may affect skin condition during the study.
  Arms: Microneedle with Saline
Drug: Microneedle with 1.2mg Denosumab — This intervention uses microneedle patches loaded with 1.2mg of denosumab. The patch is made of a biocompatible material, polyvinyl pyrrolidone (PVP), and is applied to the skin around the knee. It aims to evaluate the skin safety and tolerability of the microneedle patch at this specific dose. Participants will apply 4 microneedle patches around their knee and avoid behaviors that may affect skin condition during the study.
  Arms: Microneedle with 1.2mg Denosumab
Drug: Microneedle with 6mg Denosumab — This intervention uses microneedle patches loaded with 6mg of denosumab. The patch is made of a biocompatible material, polyvinyl pyrrolidone (PVP), and is applied to the skin around the knee. It aims to evaluate the skin safety and tolerability of the microneedle patch at this specific dose. Participants will apply 4 microneedle patches around their knee and avoid behaviors that may affect skin condition during the study.
  Arms: Microneedle with 6mg Denosumab

SUMMARY:
The goal of this clinical trial is to evaluate the skin safety of a soluble denosumab microneedle patch in participants with osteoporosis and osteoarthritis. The main questions it aims to answer are:

* Is the soluble denosumab microneedle patch safe for use on the skin?
* What are the potential skin reactions to the patch?

Researchers will compare different doses of the microneedle patch to assess its safety.

Participants will:

* Apply the microneedle patch to four different areas around their knee
* Undergo skin assessments at various time points after application
* Be monitored for any adverse skin reactions

The study will take place at a single center and involve a small number of participants to provide preliminary data on the safety of this novel drug delivery system.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent.
2. Commitment to comply with the study protocol and cooperate throughout the study.
3. Age 18-70, healthy or adult male or female with osteoarthritis combined with osteoporosis.
4. No history of skin diseases or other underlying conditions.
5. No antihistamines, vasodilators, vasoconstrictors, anticoagulants, hormones, or immunosuppressants within the past month.
6. If of childbearing age, women must have used contraception for at least one month before screening and commit to using contraception throughout the study period and for a specified time after the study ends.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Smoking >10 cigarettes per day or smoking history >20 years.
3. Presence of conditions that may interfere with the study results (e.g., severe diseases, infectious diseases, allergies, etc.) or relevant medical history.
4. Individuals receiving systemic or local treatments that affect skin homeostasis.
5. Allergic or intolerant to polyvinylpyrrolidone (PVP) or polyvinyl alcohol (PVA).
6. Contraindications for denosumab (e.g., hypocalcemia).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Reactions | Assessed at 15 minutes, 24 hours, 48 hours, and 2 weeks post-application.
  Evaluate through skin response sheets: erythema, pain, swelling, etc.
Amount of pain | Assessed at 15 minutes, 24 hours, 48 hours, and 2 weeks post-application.
  Pain will be measured using the faces pain scales revised (0-2-4-6-8-10, 0: no pain, 10: very much pain).
Number of injection site reactions | Assessed at 15 minutes, 24 hours, 48 hours, and 2 weeks post-application.
  Injection site assessment for the following:
  Pain (grade 1/2/3) Tenderness (grade 1/2/3) Pruritus (grade 1/2/3) Erythema (absent/present) Induration (grade 1/2/3) Blister (absent/present) Ulceration (absent/present) Necrosis (absent/present) Ecchymosis (absent/present) If any of these signs or symptoms is present, it is regarded an injection site reaction.

SECONDARY OUTCOMES:
Soluble Denosumab Microneedle Patch Subject Satisfaction Questionnaire | Assessed at 2 weeks post-application.
  Assessed through questionnaires at the end of the study.
  1. How satisfied are you with the application process of the microneedle patch?
  2. How satisfied are you with the overall skin condition around the knee after using the microneedle patch?
  3. Overall, how satisfied are you with the ease of using the microneedle patch?
  4. Overall, now that you have tried this microneedle patch and completed the study, how likely are you to use this treatment again in the future?
  5. Overall, how likely are you to recommend this microneedle patch treatment to a family member or friend? 5 = Very Likely; 4 = Somewhat Likely; 3 = Neutral; 2 = Somewhat Unlikely; 1 = Very Unlikely
Number of participants with abnormal laboratory tests results | Assessed at 2 weeks post-application.
  Evaluation of blood routine and blood electrolytes to monitor participants' health status and safety.

OTHER OUTCOMES:
Frequency of both local and systemic Adverse Events | 2 weeks
  An adverse event is any adverse change from the subject's baseline condition, i.e. any subjective signs and symptoms, or change in a concomitant disease present at the screening visit. This includes inter-current signs, symptoms, illness and significant deviations from baseline which may occur during the course of the clinical study, whether considered related to treatment or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT07085520/Prot_SAP_000.pdf